CLINICAL TRIAL: NCT01173653
Title: A Randomized Controlled Trial of Directed Smoking Cessation Intervention in the Emergency Care Population
Brief Title: Smoking Cessation Invention in the Emergency Department (ED)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Ben Heavrin, Benjamin S. Heavrin, MD, MBA, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 100411
Record Dates: First submitted 2010-07-29; First posted 2010-08-02 (Estimated); Results first posted 2012-11-19 (Estimated); Last update posted 2012-12-27 (Estimated); Status verified 2012-12

CONDITIONS: Smoking Cessation; Tobacco Use Cessation; Health Behavior
Keywords: smoking; smoking cessation; health behavior
MeSH Terms: conditions — Smoking Cessation; Tobacco Use Cessation; Health Behavior; Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard EM Smoking Cessation Info (Placebo Comparator): Patients discharged from ER receive pamphlet re: smoking cessation
  Interventions: Other: Smoking Cessation
- Patients contact 1-800-QUIT-NOW before leaving ED (Active Comparator): Prior the patient leaving the ED, the PI will assist the patient with contacting 1-800-QUIT-NOW, who will help patient to quit smoking.
  Interventions: Other: Smoking Cessation

INTERVENTIONS:
Other: Smoking Cessation — Randomly introducing patients to a Department of Health program to help them quit smoking.
  Arms: Standard EM Smoking Cessation Info
Other: Smoking Cessation — A simple intervention where ED patients who were motivated to quit smoking were put in direct phone contact with a trained smoking cessation counselor during their ED stay.
  Arms: Patients contact 1-800-QUIT-NOW before leaving ED

SUMMARY:
The emergency department (ED) serves a vital and growing role in the US health care system, responsible for both the delivery of emergent medical care and for safety-net care for populations without traditional access to health services. Uninsured populations rely significantly on the safety-net services of the ED. Between 2000-2005 the number of uninsured Americans increased from 39.6 million to 46.1 million, and this growth is expected to continue. Many health policy analysts consider the ED to be an effective place to provide preventative care. Prophylactic tetanus immunization, for example, has been a successful preventive health intervention that has become a standard of care in the ED setting. Brief smoking cessation interventions have been introduced in the ED but have not had great success based on lack of follow-up and continuity.

Our study is novel in that it introduces a brief smoking intervention through use of an established, federally-funded and federally-sponsored cessation counseling resource, the National Smoking Cessation Quit Line, also available at smokefree.gov. This is a joint initiative between the Tobacco Control Research Branch of the National Cancer Institute and the Centers for Disease Control and Prevention. Since ED patients who smoke often lack the ability to use self-help cessation resources, we hypothesize that by introducing this population to the counselors on the National Smoking Cessation Quit Line (also called the 1-800-QUIT-NOW line) during the ED visit via phone, that this new brief intervention would have a realizable and significant effect on smoking cessation among the this population.

DETAILED DESCRIPTION:
Smoking is a public health epidemic. Over 20% of adults in the USA smoke according to the American Heart Association. Benefits of smoking cessation are realizable and readily apparent: reductions in the risk of heart, kidney, and lung disease, reduction in the risk of stroke and certain cancers, blood pressure improvement, increased life expectancy, economic benefits, and the positive externality in secondhand smoke reduction are some of the more common benefits cited by public health experts. Smoking remains the leading preventable cause of chronic illness in our country, and, despite the well-publicized benefits, quitting smoking remains difficult. Many smokers do not wish to undergo the negative physiological effects of detoxification from nicotine dependence. Others lack the resources, support and motivation to make this lifestyle change. Providers, moreover, struggle to find a simple, effective intervention that will help their smoking population kick the habit.

Given this background, our research proposal has the following specific aims:

1. The ED is an effective location within the domestic health system to provide preventive medical care, including counseling on smoking cessation.
2. A simple intervention where ED patients who were motivated to quit smoking were put in direct phone contact with a trained smoking cessation counselor, during their ED stay, will have a realizable benefit in rates of smoking cessation beyond the placebo rate of cessation.
3. We hypothesize that smokers who are motivated to quit will react positively to the national quit line and will have a higher rate of cessation at two months time compared to other motivated smokers in the ED department who are not put in immediate contact with a smoking cessation counselor.

A background statistical analysis and literature review has already been conducted. A literature review has been attached for reference (see Appendix A). We have discussed this topic with our biostatistical liaison and we believe such a study can show statistical significance with appropriate power based on a target enrollment of 150 patients.

Following anticipated IRB approval, we expect this study to be ready for enrollment. Mr. Pelster will be the lead enrollee within the Adult Emergency Department and has the full support of the ED faculty and staff for this work. He will be supervised directly by Dr. Benjamin Heavrin, Assistant Professor of Emergency Medicine, who will function as his faculty sponsor through the VUSM emphasis program. All patients presenting to the Adult Emergency Department are asked about smoking status through the triage note. Mr. Pelster will have access to this triage note and will approach patients who meet inclusion criteria. Our inclusion criteria includes: verbally consenting patients of the Adult ED who actively smoke, have normal vital signs, and are not emergency will based on triage criteria. Exclusion criteria includes patients unable to provide consent, unable to verbally communicate, patients with emergent illness defined by ESI triage protocols, patients with unstable vitals, and patients under the age of 18. Mr. Pelster will then approach these patients for possible enrollment. Prior to the beginning of this study, Mr. Pelster will become well read on current smoking statistics and on the medical and health related benefits of smoking cessation, should patient questions arise. He will be supervised in these verbal patient discussions by Dr. Heavrin.

All patients will be asked for voluntary, verbal informed consent. Should consent not be given, or should consent not be able to be obtained, a patient will not be included in this study. Given that no harm could come from this intervention in the ED, and given that the "intervention" is simply a verbal discussion on the motivation to quit smoking and a telephone conversation with a 1-800-QUIT-NOW professional, we believe that verbal consent would be acceptable. Patients who consent to the study will be given a letter that briefly explains the purpose of the clinical trial (see Appendix B).

Basic demographic data related to age, gender, race, smoking history, and contact information of the patient will be collected and stored on a secure electronic device as described below. Upon conclusion of enrollment, data analysis will begin using statistical software such as SPSS available through the Department of Emergency Medicine, Division of Research.

Although our investigative team does not have experience in smoking cessation research, plenty of evidence exists within the medical literature to suggest that studies on smoking cessation are simple in design, context, and data acquisition and that patients respond positively to preventive health interventions. Our investigative team will be working under the Division of Research, Department of Emergency Medicine, Vanderbilt University Medical Center. This department has plentiful resources to conduct this simple investigation, including biostatistical support, dedicated clinical trials associates, and a culture of rigorous and supportive academic investigation within the clinical wings of the department.

We expect no negative impact of this investigating on clinical care, the timeliness of care, or the disposition and treatment of the patients enrolled.

A literature search has been conducted and is included. Per our review, we do not believe that research into the utilization of the 1-800-QUIT-NOW line has occurred in an Adult ED population. Should our research prove our hypothesis, this would provide a simple intervention that would have large-scale positive public health ramifications for the ED smoking population.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age and older
* Patients who are active smokers who present to the Adult ED at VUMC
* Patients who are able to give informed verbal consent
* Patients with stable vital signs

Exclusion Criteria:

* Patients who are unable to provide consent
* Patients who are unable to communicate verbally as determined by the treating attending physician and/or triage nurse. This includes patients with alterations in mental status, who are cognitively impaired, or are intoxicated or on drugs
* Patients with abnormal vital signs, and triage ratings (ES1 score 1) suggesting immediate life threatening illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2010-07; Primary Completion 2010-10 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ben Heavrin, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center - Emergency Medicine, Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 199 subjects were recruited during June and July 2010. 90 subjects were randomized to the intervention arm and 109 were randomized to the control arm.
Pre-assignment Details: The targeted patient population were patients presenting to the emergency department who were smokers. There were no restrictions placed on gender, race, or ethnicity.
Period: Overall Study
Arm/Group | Standard EM Smoking Cessation Info | Patients Contact 1-800-QUIT-NOW Before Leaving ED
Started | 109 | 90
Completed | 56 | 49
Not Completed | 53 | 41
Not completed — Pts unwilling to provide follow-up | 53 | 41

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard EM Smoking Cessation Info | Patients Contact 1-800-QUIT-NOW Before Leaving ED | Total
Number analyzed (Participants) | 109 | 90 | 199
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 109 | 90 | 199
  >=65 years | 0 | 0 | 0
Age Continuous [Median (Inter-Quartile Range); unit: years] | 44 (31, 51) [31 to 51] | 44 (33, 49) [33 to 49] | 44 (33, 50) [32 to 50]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 45 | 101
  Male | 53 | 45 | 98
Region of Enrollment [Number; unit: participants]
  United States | 109 | 90 | 199

OUTCOME MEASURES:

1. Primary Outcome: Smoking Status at Follow up
Description: Patients enrolled in this study were contacted via phone to assess smoking status. Smoking status was a self-report from each subject. Primary outcome measure is the smoking status of the enrollee at the time of follow-up contact. We calculated the percentage of participants who had stopped smoking at the 6 week follow-up period in each arm
Time Frame: 6 weeks
Population: Of subjects enrolled, 56 of the 109 subjects in the control arm and 49 of 90 subjects in the intervention arm were able to be contacted via phone and were willing to provide follow-up data for analysis of smoking status at the 6 week follow-up.
Measure: Number; unit: percentage of participants
Groups:
- Control Arm: No intervention given to this ED population of smokers
- Intervention Arm: Enrollees put in contact with 1-800-QUIT-NOW line
Arm/Group | Control Arm | Intervention Arm
Number analyzed (Participants) | 56 | 49
percentage of participants | 7 | 24
Statistical Analysis 1: Comparison: Control Arm vs Intervention Arm; Test type: Superiority or Other; p < 0.05, Chi-squared; Chi square = 23.02

ADVERSE EVENTS:
Arm/Group | Standard EM Smoking Cessation Info | Patients Contact 1-800-QUIT-NOW Before Leaving ED
Serious Adverse Events (participants affected / at risk) | 0/109 | 0/90
Other Adverse Events (participants affected / at risk) | 0/109 | 0/90

LIMITATIONS AND CAVEATS:
This is a preliminary study with a convenience sample of patients at a single academic medical center. A larger multicenter trial targeting consecutive ED patients who smoke will be essential to validate the applicability of our findings.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes